CLINICAL TRIAL: NCT04757064
Title: Efficacy of Selected Exercise Program on Distal End Femoral Sarcoma Patients Undergoing Knee Modular Endoprosthesis: RCT
Brief Title: Efficacy of Exercise Program on Osteosarcoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gamila Saleh Tammam Abbas, orthopedic physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: exercises in osteosarcoma
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Intervention Model Description: Group (A) will receive the standard protocol of king Hussein hospital 6 weeks post-operative which is:
  Start aggressive knee flexion exercises and increase the extensor strength. Consider CPM/dynasplint if flexion <60_ MUA contraindicated.
  Examination under anesthesia can be done to assess the cause of limited knee flexion. Surgical release is indicated if knee flexion is < 60 degrees at six months after surgery.
  Group (B) will receive supervised rehabilitation program 1 session / week for 45 minutes-1 hour.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Rehabilitation Group (Experimental): Standard Rehabilitation Group: will receive the standard protocol of king Hussein hospital 6 weeks post-operative which is:
  Start aggressive knee flexion exercises and increase the extensor strength. Consider CPM/dynasplint if flexion <60_ MUA contraindicated.
  Examination under anesthesia can be done to assess the cause of limited knee flexion. Surgical release is indicated if knee flexion is < 60 degrees at six months after surgery.
  Interventions: Other: standard rehabilitation protocol
- Supervised Rehabilitation Group (Experimental): Supervised Rehabilitation Group: will receive supervised rehabilitation program 1 session / week for 45 minutes-1 hour.
  Interventions: Other: standard rehabilitation protocol

INTERVENTIONS:
Other: standard rehabilitation protocol — they will receive knee flexion exercises and increase the extensor strength

SUMMARY:
This study will be conducted to investigate the effect of selected therapeutic exercises compared to standard exercise program in improving ROM, muscle strength and functional outcomes in distal femur osteosarcoma patients who have undergone tumor resection and modular knee endoprosthesis.

DETAILED DESCRIPTION:
Osteosarcomas (OS) are the most common primary bone tumor and third most common cancer among children and adolescents after lymphomas and brain cancers (Wang et al., 2018; Luetke et al., 2014).

It is a primary malignant bone tumor with a worldwide incidence of 3.4 per million people per year (Mirabello et al., 2009). They are characterized by the production of osteoid, or immature bone, by malignant mesenchymal cells (Wang et al., 2018; (Luetke et al., 2014).

Patients displayed some persisting physical difficulties including incapability to perform active range of motion (ROM), decreased muscle strength, altered gait and sit-to-stand patterns, yet they maintained high levels of emotional acceptance and coping. A surprising but important finding was the persisting hip weakness in both operated and non-operated limbs, which extends up to 42 months after resection around the knee. This indicates that continued rehabilitation programs emphasizing hip strengthening should be considered for these patients, even years after surgery (Beebe et al., 2009). Furthermore, ROM exercises, strengthening exercises and balance exercises improve overall Quality of life (QOL) for these patients (Marchese et al., 2006).

ELIGIBILITY:
Inclusion Criteria:

1) Patients diagnosed as distal femur osteosarcoma. 2) Age of the patient from 15-50 years old 3) Patients undergoing tumor resection and knee endoprosthetic reconstruction six weeks ago. 4) Both gender

-

Exclusion Criteria:

1) Lung and bone metastasis 2) End stage patients receiving palliative chemotherapy 3) Patients undergoing L.L amputation or rotationplasty (any surgical procedures rather than knee endoprosthetic reconstruction). 4) Local tumor recurrence 5) Sever psychiatric illness 6) Heart disease or any condition that prevent the patient from participation in exercise

-

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-07 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
ROM | 3 minutes
  knee flexion and extension ROM measured by goniometer
knee extensor muscle strength | 5 minutes
  measuring rectus femoris muscle strength by manual muscle testing

SECONDARY OUTCOMES:
functional outcome | 2 minutes
  measurd by Musculoskeletal Tumor Society Rating Scale, minimum score is 0 and maximum score is 30 (higher scores indicating better function)

REFERENCES:
- [Background] Galvao DA, Taaffe DR, Spry N, Cormie P, Joseph D, Chambers SK, Chee R, Peddle-McIntyre CJ, Hart NH, Baumann FT, Denham J, Baker M, Newton RU. Exercise Preserves Physical Function in Prostate Cancer Patients with Bone Metastases. Med Sci Sports Exerc. 2018 Mar;50(3):393-399. doi: 10.1249/MSS.0000000000001454. PMID 29036016
- [Background] Keilani M, Kainberger F, Pataraia A, Hasenohrl T, Wagner B, Palma S, Cenik F, Crevenna R. Typical aspects in the rehabilitation of cancer patients suffering from metastatic bone disease or multiple myeloma. Wien Klin Wochenschr. 2019 Nov;131(21-22):567-575. doi: 10.1007/s00508-019-1524-3. Epub 2019 Jul 2. PMID 31267163